CLINICAL TRIAL: NCT00510211
Title: An Observational Study of Olanzapine Coated and Orodispersible Tablets Effectiveness in Schizophrenic and Bipolar Outpatients.
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 11610; F1D-FR-B035
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- olanzapine coated tablet
  Interventions: Drug: olanzapine
- olanzapine orodispersable tablet
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine

SUMMARY:
The primary objective of this study is to assess the proportion of schizophrenic patients and the proportion of bipolar patients who discontinue olanzapine within 12 months of treatment in outpatient, ambulatory or community settings

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from schizophrenic or schizoaffective disorders based on the disease diagnostic criteria DSM IV and being prescribed olanzapine during the 45 preceding days.
* patients suffering from bipolar disorders based on the disease diagnostic criteria DSM IV and being prescribed olanzapine during the 45 preceding days for one of the following:
* moderate or severe manic episode
* relapse prevention in patients with bipolar disorder

Exclusion Criteria:

* current treatment with any investigational drug or procedure at entry or during the whole study
* hypersensitivity to olanzapine
* patients with known narrow angle glaucoma risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients observed in outpatient settings (ambulatory and community)
Sampling Method: Non-Probability Sample
Enrollment: 1131 (Actual)
Dates: Start 2007-04; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-615-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Homburg, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki, Greece

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://lillytrials.com